CLINICAL TRIAL: NCT01378858
Title: Varenicline Smoking Cessation Treatment for Methadone Maintenance Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shadi Nahvi, Assistant Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-279; K23DA025736 (NIH)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Tobacco Use Disorder; Medication Adherence
Keywords: Smoking; Substance-Related Disorders; medication adherence; Methadone
MeSH Terms: conditions — Tobacco Use Disorder; Medication Adherence; Smoking; Substance-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline treatment as usual (TAU) (Experimental): Subjects in the TAU arm will self administer varenicline for 12 weeks.
  Interventions: Drug: Varenicline
- Varenicline directly observed therapy (Experimental): Subjects in the directly observed therapy (DOT) arm will receive varenicline directly administered by methadone clinic nurses 4-6 times per week at the same time as they receive methadone, as well as individually packaged take-home doses for self administration on evenings/weekends.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline, titrated to 1 mg twice daily, will be given to participants in both study arms for 12 weeks.
  Other Names: Chantix

SUMMARY:
This randomized trial will evaluate whether varenicline directly observed therapy provided at a methadone clinic is more efficacious than self-administered varenicline for promoting smoking cessation and enhancing adherence.

DETAILED DESCRIPTION:
There is a marked prevalence of tobacco use and tobacco-related disease among methadone maintenance patients. Varenicline's demonstrated efficacy may not be generalizable to methadone maintained smokers because of poor adherence, which is highly prevalent among drug users. Adherence to smoking cessation medication is strongly associated with cessation, and is one of the few factors shown to increase cessation among methadone maintained smokers, but strategies to promote smoking cessation medication adherence have not been evaluated in methadone patients. Based on the Information, Motivation, and Behavior model, the investigators plan a directly observed therapy (DOT)-based intervention targeting behavioral skills necessary for optimal adherence. Because methadone clinic-based DOT interventions have been shown to improve medication adherence and clinical outcomes in HIV and TB, the investigators plan to determine in a randomized trial whether DOT varenicline provided at a methadone clinic is more efficacious than self-administered varenicline for promoting smoking cessation and enhancing adherence. The investigators will also evaluate moderating effects of drug and alcohol use and psychiatric symptoms on DOT effects. The investigators hypothesize subjects in the mDOT arm will have greater 7 day point prevalence abstinence at 12 weeks, reduction in cigarettes/day, time to first daily cigarette, ≥ 24 hour quit attempts, and 7 day point prevalence abstinence at 24 weeks compared to subjects receiving self administered varenicline. The investigators also hypothesize that adherence in the mDOT arm will be higher than in the TAU arm. Lastly the investigators hypothesize that ongoing illicit drug use and psychiatric symptoms will moderate the effect of mDOT on adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* English speaking
* Smoked at least 100 cigarettes/lifetime
* Smoke 5 or more cigarettes per day
* Interested in quitting smoking (preparation or contemplation stage of change)
* Enrolled in Einstein/Montefiore methadone program for 12 weeks or more
* Receiving methadone in clinic three, four, five or six times per week
* No more than 2 methadone clinic misses in prior 14 days
* Agree to use contraception for the duration of the trial (among women with reproductive potential)
* Willing to participate in all study components
* Able to provide informed consent

Exclusion Criteria:

* Serious or unstable HIV/AIDS, liver, cardiovascular, or pulmonary disease
* Psychiatric instability
* Women who are pregnant, breastfeeding, or contemplating pregnancy
* Creatinine clearance <30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Nahvi, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Nahvi S, Adams TR, Ning Y, Zhang C, Arnsten JH. Effect of varenicline directly observed therapy versus varenicline self-administered therapy on varenicline adherence and smoking cessation in methadone-maintained smokers: a randomized controlled trial. Addiction. 2021 Apr;116(4):902-913. doi: 10.1111/add.15240. Epub 2020 Oct 13. PMID 32857445
- [Derived] Nahvi S, Segal KS, Litwin AH, Arnsten JH. Rationale and design of a randomized controlled trial of varenicline directly observed therapy delivered in methadone clinics. Addict Sci Clin Pract. 2014 Jun 13;9(1):9. doi: 10.1186/1940-0640-9-9. PMID 24928218

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy
Started | 50 | 50
Completed | 46 | 46
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [45 to 52] | 49 [46 to 53] | 49 [45 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 30 | 26 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 22 | 22 | 44
  Black | 13 | 17 | 30
  Mutliracial/multiethnic | 6 | 4 | 10
  White | 7 | 7 | 14
  Other | 2 | 0 | 2
Cigarettes smoked per day [Median (Inter-Quartile Range); unit: cigarettes smoked per day] | 10 [8 to 15] | 12 [8 to 20] | 10 [8 to 20]
Expired carbon monoxide [Median (Inter-Quartile Range); unit: parts per million] — A measure of the amount of carbon monoxide on a person's breath, which is checked using a Smokerlyzer monitor (Bedfont Scientific).
  parts per million | 7 [5 to 10] | 8 [5 to 10] | 7 [5 to 10]
Fagerstrom Test of Nicotine Dependence score [Median (Inter-Quartile Range); unit: units on a scale] — In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 5 [4 to 6] | 5 [4 to 7] | 5 [4 to 6]
Ladder of change score [Median (Inter-Quartile Range); unit: units on a scale] — The Ladder is a continuous measure of motivation to change smoking where a score of 1 indicates low readiness to quit smoking and a score of 10 indicates high readiness to quit smoking.
  units on a scale | 8 [7 to 8] | 8 [6 to 8] | 8 [6 to 8]
Quit importance [Median (Inter-Quartile Range); unit: units on a scale] — Quit importance measures importance of quitting smoking for participants on a scale from 1 to 10 where 1 is not important and 10 is highly important
  units on a scale | 10 [9 to 10] | 10 [9 to 10] | 10 [9 to 10]
Quit confidence [Median (Inter-Quartile Range); unit: units on a scale] — Quit confidence measures confidence in quitting smoking for participants on a scale from 1 to 10 where 1 is not confident at all and 10 is highly confident
  units on a scale | 7 [5 to 10] | 8 [6 to 10] | 8 [5 to 10]
Any past quit attempts [Number; unit: participants] | 39 | 42 | 81
Preferred brand of cigarettes menthol [Count of Participants; unit: Participants] | 46 | 42 | 88
Number of participants with unstable housing [Number; unit: participants] — Living in a shelter, temporary housing, hotel/motel, or on the street
  participants | 27 | 37 | 64
Number of participants currently employed [Count of Participants; unit: Participants] | 10 | 10 | 20
Number of participants married or living with a partner [Count of Participants; unit: Participants] | 19 | 26 | 45
Lifetime major depressive episode [Count of Participants; unit: Participants] — Assessed using the Mini-International Neuropsychiatric Interview 6.0.0. The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a short structured diagnostic interview for assessing DSM-IV and ICD-10 psychiatric disorders.
  Participants | 10 | 11 | 21
Lifetime psychotic disorder [Count of Participants; unit: Participants] — Assessed using the Mini-International Neuropsychiatric Interview 6.0.0. The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a short structured diagnostic interview for assessing DSM-IV and ICD-10 psychiatric disorders.
  Participants | 6 | 4 | 10
Lifetime suicide attempt [Count of Participants; unit: Participants] — Assessed using the Columbia Suicide Severity Scale, a structured interview which assesses suicidal ideation, plans, intent, and behavior
  Participants | 7 | 8 | 15
Severe global psychiatric symptoms [Count of Participants; unit: Participants] — Assessed using the Brief Symptom Inventory Global Severity Index, a 53-item self report scale, with scores dichotomized at a T score ≥ 63
  Participants | 8 | 9 | 17
Currently receiving psychiatric treatment [Count of Participants; unit: Participants] | 19 | 18 | 37
Participants with COPD/Asthma [Count of Participants; unit: Participants] | 15 | 15 | 30
Participants with HIV/AIDS [Count of Participants; unit: Participants] | 9 | 11 | 20
Median duration methadone maintenance [Median (Inter-Quartile Range); unit: years] | 5 [3.3 to 8.9] | 5.6 [3.3 to 8.9] | 5.6 [3.3 to 8.9]
Median methadone dose [Median (Inter-Quartile Range); unit: mg] | 92 [60 to 120] | 83.5 [70 to 110] | 90 [61.5 to 112.5]

OUTCOME MEASURES:

1. Primary Outcome: Varenicline Adherence as Measured by Pill Count
Description: Pill count adherence, measured as pills taken divided by pills dispensed, analyzed as a continuous measure
Time Frame: Weeks 0-1, 1-2, 2-3, 4-6, 7-9, 10-12
Population: Comparison of varenicline TAU and DOT groups
Measure: Mean (95% Confidence Interval); unit: percentage pills taken/pills dispensed
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy
Number analyzed (Participants) | 50 | 50
percentage pills taken/pills dispensed | 61.8 [55.0 to 68.6] | 78.5 [71.8 to 85.2]

2. Secondary Outcome: Tobacco Abstinence Biochemically Verified With Expired Carbon Monoxide (CO) < 8 p.p.m. at 12 Weeks
Description: Number of participants achieving self reported, seven day point prevalence abstinence, biochemically verified with expired carbon monoxide (CO) < 8 p.p.m., missing = smoking
Time Frame: Week 12 of treatment
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy
Number analyzed (Participants) | 50 | 50
Participants | 9 | 5

3. Secondary Outcome: Tobacco Abstinence Biochemically Verified With Expired Carbon Monoxide (CO) < 8 p.p.m. at 24 Weeks
Description: Number of participants achieving self reported, seven day point prevalence abstinence, biochemically verified with expired carbon monoxide (CO) < 8 p.p.m.
Time Frame: 24 weeks
Population: Missing = smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy
Number analyzed (Participants) | 50 | 50
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: 12 week intervention period, and 12 week post intervention follow up
Arm/Group | Varenicline Treatment as Usual (TAU) | Varenicline Directly Observed Therapy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50 | 3/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Treatment as Usual (TAU) (N=50) | Varenicline Directly Observed Therapy (N=50)
Incident major depressive episode (Psychiatric disorders) | 0 (0) | 2 (2) — Assessed using the Mini-International Neuropsychiatric Interview 6.0.0
Incident psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) — Assessed using the Mini-International Neuropsychiatric Interview 6.0.0
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) — Wishes to be dead, or thoughts of killing self, assessed using the Columbia Suicide Severity Scale
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline Treatment as Usual (TAU) (N=50) | Varenicline Directly Observed Therapy (N=50)
Change in taste (General disorders) | 11 | 15 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Dry mouth (General disorders) | 20 | 24 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Change in appetite (General disorders) | 18 | 19 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Nausea (General disorders) | 19 | 27 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Vomiting (General disorders) | 5 | 13 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Gas (General disorders) | 10 | 17 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Constipation (General disorders) | 16 | 24 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Change in concentration (General disorders) | 4 | 7 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Headache (General disorders) | 12 | 13 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Fatigue (General disorders) | 4 | 12 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Insomnia (General disorders) | 18 | 14 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Dizziness (General disorders) | 5 | 4 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Irritability (General disorders) | 3 | 8 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment
Vivid/more frequent dreams (General disorders) | 11 | 16 — Assessed through structured questionnaire, assessing specific symptoms reported in varenicline clinical trials, and open-ended assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes